CLINICAL TRIAL: NCT04979533
Title: Oxygen Insufflation: How High Flow, Low Pressure Oxygen Can Replace Jet Ventilation in Appropriate Surgical Airway Cases
Brief Title: Oxygen Insufflation in Microlaryngoscopies
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Professional decision
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Hollie Sanders, Certified Registered Nurse Anesthetist, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB-300007262
Record Dates: First submitted 2021-06-29; First posted 2021-07-28 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Hypoxia
Keywords: surgery; airway; hypoxia prevention; oxygen insufflation
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Intervention Model Description: There will be a single group of participants in which all receive oxygen insufflation to see if oxygen insufflation is adequate in microlaryngoscopy airway surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Oxygen Insufflation (Experimental): Oxygen insufflation via oxygen tubing at 15 L/min
  Interventions: Device: Insufflator oxygen tubing

INTERVENTIONS:
Device: Insufflator oxygen tubing — high flow, low pressure oxygen with pressure relief valve and luer Lock connections delivered at 15 L/min through surgeon's laryngoscope.
  Other Names: Flexible Oxygen tubing

SUMMARY:
The purpose of this project is to evaluate the efficacy of oxygen insufflation (continuous oxygen flow) to keep oxygen saturation (oxygen levels measured with a pulse oximeter [finger device used in medicine]) at 90% or greater in adult patients undergoing microlaryngoscopy surgery.

DETAILED DESCRIPTION:
High flow, low pressure oxygen will be supplied in microlaryngoscopy airway surgery. These procedures are usually performed with jet ventilation (UAB) or intermittent apnea (surgery centers). Jet ventilation provides oxygenation with limited ventilation but come with high risks, such as barotrauma, pneumothorax, mucosa drying, and even death in the most severe cases. Intermittent apnea is a nuisance for the surgeon in that surgical time is often interrupted with having to place the endotracheal tube whenever the patient's oxygen saturation levels fall. The solution is oxygen insufflation, which will give extended oxygenation times for the surgeon to operate without the inherent risks associated with jet ventilation. During the procedure, oxygen tubing will be connected to the surgeon's laryngoscope instead of the jet ventilation tubing. Oxygen flows of 15 L/min will be administered through the laryngoscope to the posterior oropharynx. Endotracheal tube will be placed if oxygenation deemed insufficient due to oxygen saturations of <90%. Endotracheal tube will be intermittently placed to check and correct carbon dioxide levels.

ELIGIBILITY:
Inclusion Criteria:

* adult patients undergoing microlaryngoscopy surgery without a tracheostomy

Exclusion Criteria:

* patients who have a tracheostomy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
High flow, low pressure oxygen can increase apneic oxygenation time during airway procedures | 30-60 minutes
  15 liters per minute of oxygen will be administered to the posterior oropharynx.

SECONDARY OUTCOMES:
Degree of hypercapnia experienced by participants | 30-60 minutes
  Measurement will be taken by intermittent ventilation by placing an endotracheal tube
Participants That Maintain Adequate Oxygenation at 90% or Greater | 30-60 minutes
  Pulse oximetry will be used to measure oxygenation status

CONTACTS AND LOCATIONS:
Overall Officials: Hollie N Sanders, MSN, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: No
The oxygen saturation numbers throughout each surgery will be recorded with no personal identifying data of each patient.